CLINICAL TRIAL: NCT01687270
Title: A Phase 2, Multicenter, Open-Label Study to Investigate the Safety and Efficacy of GS-7977 and Ribavirin for 24 Weeks in Subjects With Recurrent Chronic HCV Post Liver Transplant
Brief Title: Safety and Efficacy of Sofosbuvir and Ribavirin in Adults With Recurrent Chronic Hepatitis C Virus (HCV) Post Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0126; 2012-002417-19 (EudraCT Number)
Expanded Access: NCT01779518 (Approved for marketing)
Record Dates: First submitted 2012-09-12; First posted 2012-09-18 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Recurrent Chronic Hepatitis C Virus; Post Liver Transplant
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOF+RBV (Experimental): Participants will receive sofosbuvir+RBV for 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet administered orally once daily
  Other Names: GS-7977; PSI-7977; Sovaldi®
Drug: RBV — Ribavirin (RBV) 200-mg tablet(s) administered orally in a divided daily dose starting at 400 mg, subsequently adjusted (range: 200 to 1200 mg in a divided daily dose) based upon a number of factors including hemoglobin value, creatinine clearance, and weight.
  Other Names: Ribasphere®

SUMMARY:
This is an open-label, single-arm study of sofosbuvir (GS-7977) and ribavirin (RBV) in adults who have had a liver transplant which has become re-infected with hepatitis C. The treatment period is 24 weeks with up to 48 weeks of follow up. The total time in this study will last up to 72 weeks not including the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with evidence of chronic HCV (all genotypes) documented pretransplantation
* HCV RNA ≥ 10,000 IU/mL at screening
* Absence of organ rejection as documented by post transplant liver biopsy taken no more than 12 months prior to baseline/Day 1 visit
* Liver transplant ≥ 6 months and ≤ 12 years prior to screening
* Naive to all nucleotide/nucleoside treatments for chronic HCV infection

Exclusion Criteria:

* Multiorgan transplant that includes heart or lung recipient
* Subjects with de novo or recurrent Hepatocellular Carcinoma(HCC) post transplant
* Current use of corticosteroids at any dose > 5mg of prednisone/day (or equivalent dose of corticosteroid)
* Infection with hepatitis B virus (HBV) or HIV at screening
* Current, uncontrolled ascites, variceal hemorrhage, hepatic encephalopathy, hepatorenal syndrome, hepatopulmonary syndrome, or other signs of decompensated cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M. Denning, MA, Study Director — Gilead Sciences
Locations (11):
- United States (7):
  - San Francisco, California
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - New York, New York
- Villejuif, France
- Hanover, Lower Saxony, Germany
- Grafton, Auckland, New Zealand
- Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Charlton M, Gane E, Manns MP, Brown RS Jr, Curry MP, Kwo PY, Fontana RJ, Gilroy R, Teperman L, Muir AJ, McHutchison JG, Symonds WT, Brainard D, Kirby B, Dvory-Sobol H, Denning J, Arterburn S, Samuel D, Forns X, Terrault NA. Sofosbuvir and ribavirin for treatment of compensated recurrent hepatitis C virus infection after liver transplantation. Gastroenterology. 2015 Jan;148(1):108-17. doi: 10.1053/j.gastro.2014.10.001. Epub 2014 Oct 7. PMID 25304641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 12 study sites in the United States, Europe, and New Zealand. The first participant was screened on 26 October 2012. The last participant observation occurred on 14 August 2014.
Pre-assignment Details: 49 participants were screened.
Groups:
- SOF+RBV: Sofosbuvir (SOF) 400 mg tablet once daily plus ribavirin (RBV) tablets (400 mg daily starting dose, then adjusted to 200-1200 mg daily) for 24 weeks
Period: Overall Study
Arm/Group | SOF+RBV
Started | 40
Completed | 28
Not Completed | 12
Not completed — Lack of Efficacy | 11
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were enrolled and received at least one dose of study medication.
Groups:
- SOF+RBV: SOF 400 mg tablet once daily plus RBV tablets (400 mg daily starting dose, then adjusted to 200-1200 mg daily) for 24 weeks
Arm/Group | SOF+RBV
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 34
  Black | 3
  Asian | 2
  Other | 1
Region of Enrollment [Number; unit: participants]
  France | 3
  United States | 28
  Spain | 3
  Germany | 3
  New Zealand | 3
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.55 (0.751)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 8
  6 to 7 log10 IU/mL | 20
  > 7 log10 IU/mL | 12
Prior HCV Treatment [Number; unit: participants]
  No | 5
  Yes | 35
HCV Genotype [Number; unit: participants]
  Genotype 1A | 22
  Genotype 1B | 11
  Genotype 3A | 5
  Genotype 3B | 1
  Genotype 4 | 1
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 13
    CT | 16
    TT | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, < 25 IU/mL) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants were enrolled and received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 40
percentage of participants | 70.0

2. Primary Outcome: Percentage of Participants Who Discontinue Study Drug Due to an Adverse Event
Time Frame: Baseline to Week 24
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 40
percentage of participants | 5.0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 4, 24, and 48 Weeks After Discontinuation of Therapy (SVR4, SVR24, and SVR48)
Description: SVR4, SVR 24, and SVR 48 were defined as HCV RNA < LLOQ 4, 24, and 48 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4, 24, and 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 40
percentage of participants
  SVR4 | 72.5
  SVR24 | 70.0
  SVR48 | 70.0

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 12 and 24
Time Frame: Weeks 12 and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 40
percentage of participants
  Week 12 (n = 40) | 100.00
  Week 24 (n = 38) | 100.00

5. Secondary Outcome: HCV RNA and Change From Baseline at Weeks 2, 4, and 8
Time Frame: Baseline; Weeks 2, 4, and 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV
Number analyzed (Participants) | 40
log10 IU/mL
  Week 2 (n = 39) | 1.65 (0.370)
  Change from baseline at Week 2 (n = 39) | -4.89 (0.692)
  Week 4 (n = 40) | 1.38 (0.000)
  Change from baseline at Week 4 (n = 40) | -5.17 (0.751)
  Week 8 (n = 40) | 1.38 (0.005)
  Change from baseline at Week 8 (n = 40) | -5.17 (0.752)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as on-treatment virologic failure or virologic relapse.
  * On-treatment virologic failure: HCV RNA < LLOQ during treatment with subsequent detectable HCV RNA while continuing treatment
  * Virologic relapse: HCV RNA < LLOQ at last observed on-treatment HCV RNA measurement and HCV RNA ≥ LLOQ after stopping treatment (2 consecutive HCV RNA measurements or last available HCV RNA measurement)
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 40
percentage of participants
  On-treatment virologic failure | 0
  Virologic relapse | 30.0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis set
Arm/Group | SOF+RBV
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=40)
Ascites (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Jaundice (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=40)
Anaemia (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 4
Oral lichen planus (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 12
Asthenia (General disorders) | 4
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 3
Candida infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 2
Blood creatinine increased (Investigations) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Irritability (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years